CLINICAL TRIAL: NCT02807038
Title: Longitudinal Study of the Pulmonary Function Testing of Pregnant Women Exposed to Air Pollution in São Paulo
Brief Title: Assessment of Exposures of the Mother-infant Pair to the Air Pollution of São Paulo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0205.0162.162-10
Record Dates: First submitted 2016-06-08; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2014-11

CONDITIONS: Lung Diseases
Keywords: Respiratory Function Tests; Air pollution; Pregnancy; Spirometry
MeSH Terms: conditions — Lung Diseases | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lung function test (Experimental): Pregnant women performed one spirometry at each trimester of pregnancy
  Interventions: Procedure: Lung function test

INTERVENTIONS:
Procedure: Lung function test — Pregnant woman use the individual passive sampler 15 days before the spirometry test at each trimester
  Other Names: Spirometry

SUMMARY:
A single group of pregnant women who was analyzed in the first and in the third trimesters of pregnancy

DETAILED DESCRIPTION:
A single group of 120 pregnant women separated in smokers (n = 17) and nonsmokers (n = 103) and first pregnancy (n = 54) or multiparous (n = 66) who underwent pulmonary function test and used the individual passive sampler in the first and third trimesters of pregnancy

ELIGIBILITY:
Inclusion Criteria:

* prior informed consent;
* single pregnancy;
* topical and feasible;
* gestational age of less than 13.86 weeks at the first evaluation;
* absence of preexisting maternal diseases

Exclusion Criteria:

* withdrawal from the project;
* abortion;
* inadequate pulmonary function test

Ages: 15 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Effect of air pollution in the spirometry of 120 pregnants, evaluated by individual passive samplers in the first (T1) and third (T3) trimesters of pregnancy, using the non-parametric analysis for repeated measures | Through study completion, an average of 3 year

SECONDARY OUTCOMES:
Evaluation of the influence of smoking and parity and the results of spirometry of all pregnants exposed to pollution comparing the frequency of events held by Wilcoxon and the Mann Witney test | Through study completion, an average of 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Duzolina M Pastro, PhD, Principal Investigator — School of Medicine, University of São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pastro LDM, Lemos M, Fernandes FLA, Saldiva SRDM, Vieira SE, Romanholo BMS, Saldiva PHN, Francisco RPV. Longitudinal study of lung function in pregnant women: Influence of parity and smoking. Clinics (Sao Paulo). 2017 Oct;72(10):595-599. doi: 10.6061/clinics/2017(10)02. PMID 29160421